CLINICAL TRIAL: NCT01681186
Title: A Single Ascending Dose and Relative Bioavailability Study of LY2940680 in Healthy Subjects
Brief Title: A Study of LY2940680 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 14893; I4J-MC-HHBG (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-09

CONDITIONS: Healthy Participants
MeSH Terms: interventions — LY2940680; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- LY2940680 (Part A) (Experimental): Single escalating dose (50 mg up to 400 mg) of LY2940680 given once orally in up to 2 of 2 study periods
  Interventions: Drug: LY2940680 Capsule(s) (Reference)
- Placebo (Part A) (Placebo Comparator): Placebo given once orally in up to 1 of 2 study periods
  Interventions: Drug: Placebo Capsule(s)
- LY2940680 Capsule Fasted (Part B) (Experimental): 100 mg LY2940680 given once orally as a capsule (reference formulation) in fasted state in 1 of 4 study periods
  Interventions: Drug: LY2940680 Capsule(s) (Reference)
- LY2940680 Tablet Fasted (Part B) (Experimental): 100 mg LY2940680 given once orally as a tablet (test formulation) in fasted state in 1 of 4 study periods
  Interventions: Drug: LY2940680 Tablet (Test)
- LY2940680 Tablet Fed (Part B) (Experimental): 100 mg LY2940680 given once orally as a tablet (test formulation) in fed state following a standardized, high-fat breakfast in 1 of 4 study periods
  Interventions: Drug: LY2940680 Tablet (Test)
- LY2940680 Tablet Fasted + PPI (Part B) (Experimental): 30 mg lansoprazole (PPI) given orally once daily for 7 days. One hour after last dose, 100 mg LY2940680 given orally once as a tablet (test formulation) in fasted state in 1 of 4 study periods
  Interventions: Drug: LY2940680 Tablet (Test); Drug: Lansoprazole

INTERVENTIONS:
Drug: LY2940680 Capsule(s) (Reference) — Administered orally as a capsule(s)
  Arms: LY2940680 (Part A); LY2940680 Capsule Fasted (Part B)
Drug: LY2940680 Tablet (Test) — Administered orally as a tablet
  Arms: LY2940680 Tablet Fasted (Part B); LY2940680 Tablet Fasted + PPI (Part B); LY2940680 Tablet Fed (Part B)
Drug: Lansoprazole — Administered orally as a capsule
  Arms: LY2940680 Tablet Fasted + PPI (Part B)
Drug: Placebo Capsule(s) — Administered orally as a capsule(s)
  Arms: Placebo (Part A)

SUMMARY:
This study involves 2 parts, Part A and Part B. The purpose of Part A is to evaluate the safety and side effects of LY2940680 in healthy participants. Part A will involve two groups of participants, each taking up to two single doses of LY2940680 at different dose levels. There is a minimum 14 day washout period between each of the participant's doses. The purpose of Part B is to study how much of the study drug, in capsule or tablet form, gets into the bloodstream and how long the body takes to get rid of it. In addition, the effect of food and a proton pump inhibitor (PPI) on LY2940680 will be studied. Part B will involve one group of participants who will take four single doses of 100 milligrams (mg) LY2940680. There is a minimum 7 day washout period between doses. Participants may only enroll in one part. Screening is required within 28 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy sterile males or surgically sterile females or postmenopausal females, as determined by medical history and physical examination
* Body mass index of 18.5 to 32.0 kilograms per meter square (kg/m^2)
* Have clinical laboratory test results within normal reference range
* Have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site
* Prepared to eat an entire high fat breakfast

Exclusion Criteria:

* Are currently enrolled in, have completed or discontinued within the last 30 days from a clinical trial involving an investigational product
* Have known allergies to LY2940680, related compounds or any components of the formulation, or known allergies to lansoprazole (Part B only)
* Have previously completed or withdrawn from this study or any other study investigating LY2940680, and have previously received the investigational product. Participants in Part A are not allowed to participate in Part B
* Have an abnormality in the 12-lead electrocardiogram (ECG)
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data (cholecystectomy or appendectomy are allowed if surgery at least 6 months prior to screening)
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Have used or intend to use over-the-counter or prescription medication within 14 days prior to dosing or during the study. Exception: participants may continue hormone replacement therapy (HRT; estrogen)
* Use of herbal supplements, grapefruit juice, grapefruits, Seville orange juice, Seville oranges, or Starfruit within 7 days prior to dosing or during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This randomized single-dose study consisted of 2 parts. Part A had Cohorts 1 and 2 receive ascending doses of LY2940680 and placebo over 2 periods. Part B had Cohort 3 receive 1 of 2 treatment sequences over 4 separate periods to evaluate tablet versus capsule (reference) formulation, and the effects of food and proton pump inhibitor (PPI).
Groups:
- Part A, Cohort 1, Sequence 1: 50-milligram (mg) LY2940680 capsule in fasted state in Period 1 followed by 200-mg LY2940680 capsule in fasted state in Period 2. There was a washout period of at least 14 days between doses in Part A of the study.
- Part A, Cohort 1, Sequence 2: 50-mg LY2940680 capsule in fasted state in Period 1 followed by Placebo in fasted state in Period 2. There was a washout period of at least 14 days between doses in Part A of the study.
- Part A, Cohort 1, Sequence 3: Placebo in fasted state in Period 1 followed by 200-mg LY2940680 capsule in fasted state in Period 2. There was a washout period of at least 14 days between doses in Part A of the study.
- Part A, Cohort 2, Sequence 4: 100-mg LY2940680 capsule in fasted state in Period 1 followed by 400-mg LY2940680 capsule in fasted state in Period 2. There was a washout period of at least 14 days between doses in Part A of the study.
- Part A, Cohort 2, Sequence 5: 100-mg LY2940680 capsule in fasted state in Period 1 followed by Placebo in fasted state in Period 2. There was a washout period of at least 14 days between doses in Part A of the study.
- Part A, Cohort 2, Sequence 6: Placebo in fasted state in Period 1 followed by 400-mg LY2940680 capsule in fasted state in Period 2. There was a washout period of at least 14 days between doses in Part A of the study.
- Part B, Cohort 3, Sequence 1: 100-mg LY2940680 capsule in fasted state in Period 1, then100-mg LY2940680 tablet in fasted state in Period 2, then 100-mg LY2940680 tablet in fed state following standardized, high-fat breakfast in Period 3, and then 100-mg LY2940680 tablet and 30-mg lansoprazole capsule in fasted state in Period 4. There was a washout period of at least 7 days between doses in Part B of the study.
- Part B, Cohort 3, Sequence 2: 100-mg LY2940680 tablet in fasted state in Period 1, then 100-mg LY2940680 capsule in fasted state in Period 2, then 100-mg LY2940680 tablet in fed state following standardized, high-fat breakfast in Period 3, and then 100-mg LY2940680 tablet and 30-mg lansoprazole capsule in fasted state in Period 4. There was a washout period of at least 7 days between doses in Part B of the study.
Period: First Intervention
Arm/Group | Part A, Cohort 1, Sequence 1 | Part A, Cohort 1, Sequence 2 | Part A, Cohort 1, Sequence 3 | Part A, Cohort 2, Sequence 4 | Part A, Cohort 2, Sequence 5 | Part A, Cohort 2, Sequence 6 | Part B, Cohort 3, Sequence 1 | Part B, Cohort 3, Sequence 2
Started | 4 | 2 | 2 | 3 | 3 | 2 | 7 | 7
Completed | 4 | 2 | 2 | 3 | 3 | 2 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period From First Intervention
Arm/Group | Part A, Cohort 1, Sequence 1 | Part A, Cohort 1, Sequence 2 | Part A, Cohort 1, Sequence 3 | Part A, Cohort 2, Sequence 4 | Part A, Cohort 2, Sequence 5 | Part A, Cohort 2, Sequence 6 | Part B, Cohort 3, Sequence 1 | Part B, Cohort 3, Sequence 2
Started | 4 | 2 | 2 | 3 | 3 | 2 | 7 | 7
Completed | 4 | 2 | 2 | 3 | 3 | 2 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Part A, Cohort 1, Sequence 1 | Part A, Cohort 1, Sequence 2 | Part A, Cohort 1, Sequence 3 | Part A, Cohort 2, Sequence 4 | Part A, Cohort 2, Sequence 5 | Part A, Cohort 2, Sequence 6 | Part B, Cohort 3, Sequence 1 | Part B, Cohort 3, Sequence 2
Started | 4 | 2 | 2 | 3 | 3 | 2 | 7 | 7
Completed | 4 | 2 | 2 | 3 | 3 | 2 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period From Second Intervention
Arm/Group | Part A, Cohort 1, Sequence 1 | Part A, Cohort 1, Sequence 2 | Part A, Cohort 1, Sequence 3 | Part A, Cohort 2, Sequence 4 | Part A, Cohort 2, Sequence 5 | Part A, Cohort 2, Sequence 6 | Part B, Cohort 3, Sequence 1 | Part B, Cohort 3, Sequence 2
Started | 0 (Part A participants received only First Intervention and Second Intervention.) | 0 (Part A participants received only First Intervention and Second Intervention.) | 0 (Part A participants received only First Intervention and Second Intervention.) | 0 (Part A participants received only First Intervention and Second Intervention.) | 0 (Part A participants received only First Intervention and Second Intervention.) | 0 (Part A participants received only First Intervention and Second Intervention.) | 7 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Third Intervention
Arm/Group | Part A, Cohort 1, Sequence 1 | Part A, Cohort 1, Sequence 2 | Part A, Cohort 1, Sequence 3 | Part A, Cohort 2, Sequence 4 | Part A, Cohort 2, Sequence 5 | Part A, Cohort 2, Sequence 6 | Part B, Cohort 3, Sequence 1 | Part B, Cohort 3, Sequence 2
Started | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period From Third Intervention
Arm/Group | Part A, Cohort 1, Sequence 1 | Part A, Cohort 1, Sequence 2 | Part A, Cohort 1, Sequence 3 | Part A, Cohort 2, Sequence 4 | Part A, Cohort 2, Sequence 5 | Part A, Cohort 2, Sequence 6 | Part B, Cohort 3, Sequence 1 | Part B, Cohort 3, Sequence 2
Started | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Fourth Intervention
Arm/Group | Part A, Cohort 1, Sequence 1 | Part A, Cohort 1, Sequence 2 | Part A, Cohort 1, Sequence 3 | Part A, Cohort 2, Sequence 4 | Part A, Cohort 2, Sequence 5 | Part A, Cohort 2, Sequence 6 | Part B, Cohort 3, Sequence 1 | Part B, Cohort 3, Sequence 2
Started | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants in Part A and B of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A, Cohort 1, Sequence 1 | Part A, Cohort 1, Sequence 2 | Part A, Cohort 1, Sequence 3 | Part A, Cohort 2, Sequence 4 | Part A, Cohort 2, Sequence 5 | Part A, Cohort 2, Sequence 6 | Part B, Cohort 3, Sequence 1 | Part B, Cohort 3, Sequence 2 | Total
Number analyzed (Participants) | 4 | 2 | 2 | 3 | 3 | 2 | 7 | 7 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 2 | 3 | 3 | 2 | 7 | 7 | 30
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 2 | 2 | 3 | 1 | 7 | 7 | 28
  Male | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 4 | 10
  Not Hispanic or Latino | 4 | 2 | 2 | 2 | 3 | 1 | 3 | 3 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 2 | 7
  White | 3 | 1 | 2 | 2 | 1 | 2 | 5 | 5 | 21
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 2 | 2 | 3 | 3 | 2 | 7 | 7 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 1 or More Adverse Events (AEs) or Any Serious AEs
Description: Data presented are the number of participants with AEs or any serious AEs (SAEs) regardless of causality. A summary of non-serious AEs is located in the Reported Adverse Events section.
Time Frame: Baseline through study completion (up to 4 weeks in Part A and 8 weeks in Part B)
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Capsule (Fasted): Placebo capsule given once orally in fasted state during Part A of the study.
- 50-mg LY2940680 Capsule (Fasted): 50-milligram (mg) LY2940680 capsule administered once orally in fasted state during Part A of the study.
- 100-mg LY2940680 Capsule (Fasted) Part A: 100-mg LY2940680 capsule administered once orally in fasted state during Part A of the study.
- 100-mg LY2940680 Capsule (Fasted) Part B: 100-mg LY2940680 capsule administered once orally in fasted state during Part B of the study.
- 100-mg LY2940680 Tablet (Fasted): 100-mg LY2940680 tablet administered once orally in fasted state during Part B of the study.
- 100-mg LY2940680 Tablet Plus 30-mg Lansoprazole (Fasted): 100-mg LY2940680 tablet administered in fasted state with a 7-day lead-in phase of once-daily 30-mg lansoprazole [proton pump inhibitor(PPI)] followed by 100-mg LY2940680 tablet administered 1 hour after the last dose of lansoprazole during Part B of the study.
- 100-mg LY2940680 Tablet (Fed): 100-mg LY2940680 tablet administered once orally in fed state following standardized, high-fat breakfast during Part B of the study.
- 200-mg LY2940680 Capsule (Fasted): 200-mg LY2940680 capsule administered once orally in fasted state during Part A of the study.
- 400-mg LY2940680 Capsule (Fasted): 400-mg LY2940680 capsule administered once orally in fasted state during Part A of the study.
Arm/Group | Placebo Capsule (Fasted) | 50-mg LY2940680 Capsule (Fasted) | 100-mg LY2940680 Capsule (Fasted) Part A | 100-mg LY2940680 Capsule (Fasted) Part B | 100-mg LY2940680 Tablet (Fasted) | 100-mg LY2940680 Tablet Plus 30-mg Lansoprazole (Fasted) | 100-mg LY2940680 Tablet (Fed) | 200-mg LY2940680 Capsule (Fasted) | 400-mg LY2940680 Capsule (Fasted)
Number analyzed (Participants) | 9 | 6 | 6 | 14 | 14 | 11 | 12 | 6 | 5
Participants
  Adverse Events (AEs) | 2 | 3 | 4 | 6 | 5 | 3 | 5 | 3 | 3
  Serious Adverse Events (SAEs) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part B: Pharmacokinetics: Maximum Observed Concentrations (Cmax) of LY2940680 Test and Reference Formulation
Description: The Cmax of 100-milligram (mg) LY2940680 capsule (reference formulation) and 100-mg LY2940680 tablet (test formulation) in fasted and fed state, and with lansoprazole during Part B of the study.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours after administration of study drug
Population: Analysis was based on the number of randomized participants in Part B of the study with evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- 100-mg LY2940680 Capsule (Fasted): 100-milligram (mg) LY2940680 capsule administered once orally in fasted state during Part B of the study.
- 100-mg LY2940680 Tablet Plus 30-mg Lansoprazole (Fasted): 100-mg LY2940680 tablet administered in fasted state with a 7-day lead-in phase of once-daily 30-mg lansoprazole [proton pump inhibitor (PPI)] followed by 100-mg LY2940680 tablet administered 1 hour after the last dose of lansoprazole during Part B of the study.
Arm/Group | 100-mg LY2940680 Capsule (Fasted) | 100-mg LY2940680 Tablet (Fasted) | 100-mg LY2940680 Tablet (Fed) | 100-mg LY2940680 Tablet Plus 30-mg Lansoprazole (Fasted)
Number analyzed (Participants) | 14 | 14 | 11 | 10
nanograms per milliliter (ng/mL) | 879 (49.3) | 1170 (22.4) | 776 (26.3) | 1290 (47.9)

3. Secondary Outcome: Part A: Pharmacokinetics: Maximum Observed Drug Concentration (Cmax)
Description: The Cmax of LY2940680 during Part A of the study was reported.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, and 120 hours after administration of study drug
Population: Analysis was based on the number of randomized participants who received LY2940680 during Part A of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- 100-mg LY2940680 Capsule (Fasted): 100-mg LY2940680 capsule administered once orally in fasted state during Part A of the study.
Arm/Group | 50-mg LY2940680 Capsule (Fasted) | 100-mg LY2940680 Capsule (Fasted) | 200-mg LY2940680 Capsule (Fasted) | 400-mg LY2940680 Capsule (Fasted)
Number analyzed (Participants) | 6 | 6 | 6 | 5
nanograms per milliliter (ng/mL) | 622 (25.3) | 661 (68.3) | 1740 (15.6) | 3360 (32.8)

4. Secondary Outcome: Part A: Pharmacokinetics: Time to Maximum Observed Drug Concentration (Tmax)
Description: Part A: Pharmacokinetics: Time to Maximum Observed Drug Concentration (tmax)
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, and 120 hours after administration of study drug
Population: Analysis was based on the number of randomized participants who received LY2940680 during Part A of the study.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | 50-mg LY2940680 Capsule (Fasted) | 100-mg LY2940680 Capsule (Fasted) | 200-mg LY2940680 Capsule (Fasted) | 400-mg LY2940680 Capsule (Fasted)
Number analyzed (Participants) | 6 | 6 | 6 | 5
hours (h) | 1.5 [0.92 to 3.0] | 2 [2.0 to 4.03] | 2 [1.0 to 2.0] | 2 [1.0 to 3.0]

5. Secondary Outcome: Part B: Pharmacokinetics: Time to Maximum Observed Drug Concentration (Tmax)
Description: Part B: Pharmacokinetics: Time to Maximum Observed Drug Concentration (tmax)
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 hours after administration of study drug
Population: Analysis was based on the number of randomized participants who received LY2940680 and had evaluable PK data during Part B of the study.
Measure: Median (Full Range); unit: hours (h)
Groups:
- 100-mg LY2940680 Tablet (Fed): 100-mg LY2940680 tablet administered once orally in fed state during Part B of the study.
- 100-mg LY2940680 Tablet (Fasted) PPI: 100-mg LY2940680 tablet administered once orally in fasted state during Part B of the study. Participants were administered 30 mg lansoprazole (proton pump inhibitor (PPI)) once-daily (QD).
Arm/Group | 100-mg LY2940680 Capsule (Fasted) | 100-mg LY2940680 Tablet (Fasted) | 100-mg LY2940680 Tablet (Fed) | 100-mg LY2940680 Tablet (Fasted) PPI
Number analyzed (Participants) | 14 | 14 | 11 | 10
hours (h) | 1 [1 to 4] | 1.5 [1 to 4] | 3 [2 to 8] | 1 [1 to 3]

6. Secondary Outcome: Part A: Pharmacokinetics: Area Under the Curve From Time Zero to Time T, Where T is the Last Time Point With a Measurable Concentration [AUC(0-tlast)]
Description: Part A: Pharmacokinetics: Area Under the Curve from Time Zero to Time T, where T is the Last Time Point with a Measurable Concentration [AUC(0-tlast)]
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, and 120 hours after administration of study drug
Population: Analysis was based on the number of randomized participants who received LY2940680 during Part A of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Arm/Group | 50-mg LY2940680 Capsule (Fasted) | 100-mg LY2940680 Capsule (Fasted) | 200-mg LY2940680 Capsule (Fasted) | 400-mg LY2940680 Capsule (Fasted)
Number analyzed (Participants) | 6 | 6 | 6 | 5
nanograms*hours per milliliter (ng*h/mL) | 5300 (27.5) | 9440 (53.9) | 22800 (21.2) | 49300 (27.9)

7. Secondary Outcome: Part B: Pharmacokinetics: Area Under the Curve From Time Zero to Time T, Where T is the Last Time Point With a Measurable Concentration [AUC(0-tlast)]
Description: Part B: Pharmacokinetics: Area Under the Curve from Time Zero to Time T, where T is the Last Time Point with a Measurable Concentration [AUC(0-tlast)]
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 hours after administration of study drug
Population: Analysis was based on the number of randomized participants who received LY2940680 who had evaluable PK data during Part B of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Groups:
- 100-mg LY2940680 Tablet (Fasted) PPI: 100-mg LY2940680 tablet administered once orally in fasted state during Part A of the study. Participants were administered 30 mg lansoprazole (proton pump inhibitor (PPI)) once-daily (QD).
Arm/Group | 100-mg LY2940680 Capsule (Fasted) | 100-mg LY2940680 Tablet (Fasted) | 100-mg LY2940680 Tablet (Fed) | 100-mg LY2940680 Tablet (Fasted) PPI
Number analyzed (Participants) | 14 | 14 | 11 | 10
nanograms*hours per milliliter (ng*h/mL) | 9390 (41.1) | 10300 (39.9) | 11200 (37.2) | 9980 (50.1)

8. Secondary Outcome: Part A: Pharmacokinetics: Area Under the Curve From Time Zero to Infinity [AUC(0-∞)]
Description: Part A: Pharmacokinetics: Area Under the Curve From Time Zero to Infinity [AUC(0-∞)]
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, and 120 hours after administration of study drug
Population: Analysis was based on the number of randomized participants who received LY2940680 during Part A of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Arm/Group | 50-mg LY2940680 Capsule (Fasted) | 100-mg LY2940680 Capsule (Fasted) | 200-mg LY2940680 Capsule (Fasted) | 400-mg LY2940680 Capsule (Fasted)
Number analyzed (Participants) | 6 | 6 | 6 | 5
nanograms*hours per milliliter (ng*h/mL) | 5340 (27.4) | 9530 (54.0) | 23000 (21.6) | 49800 (28.3)

9. Secondary Outcome: Part B: Pharmacokinetics: Area Under the Curve From Time Zero to Infinity [AUC(0-∞)]
Description: Part B: Pharmacokinetics: Area Under the Curve From Time Zero to Infinity [AUC(0-∞)]
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 hours after administration of study drug
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Arm/Group | 100-mg LY2940680 Capsule (Fasted) | 100-mg LY2940680 Tablet (Fasted) | 100-mg LY2940680 Tablet (Fed) | 100-mg LY2940680 Tablet (Fasted) PPI
Number analyzed (Participants) | 14 | 14 | 11 | 10
nanograms*hours per milliliter (ng*h/mL) | 9460 (41.3) | 10300 (40.1) | 11300 (37.3) | 10000 (50.1)

ADVERSE EVENTS:
Groups:
- 100-mg LY2940680 Capsule (Fasted) Part A or Part B: 100-mg LY2940680 capsule administered once orally in fasted state during Part A or Part B of the study.
- 100 mg LY2940680 Tablet (Fasted): 100-mg LY2940680 tablet administered once orally in fasted state during Part B of the study.
Arm/Group | Placebo Capsule (Fasted) | 50-mg LY2940680 Capsule (Fasted) | 100-mg LY2940680 Capsule (Fasted) Part A or Part B | 100 mg LY2940680 Tablet (Fasted) | 100-mg LY2940680 Tablet Plus 30-mg Lansoprazole (Fasted) | 100-mg LY2940680 Tablet (Fed) | 200-mg LY2940680 Capsule (Fasted) | 400-mg LY2940680 Capsule (Fasted)
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/20 | 0/14 | 0/11 | 0/12 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 2/9 | 3/6 | 10/20 | 5/14 | 3/11 | 5/12 | 3/6 | 3/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo Capsule (Fasted) (N=9) | 50-mg LY2940680 Capsule (Fasted) (N=6) | 100-mg LY2940680 Capsule (Fasted) Part A or Part B (N=20) | 100 mg LY2940680 Tablet (Fasted) (N=14) | 100-mg LY2940680 Tablet Plus 30-mg Lansoprazole (Fasted) (N=11) | 100-mg LY2940680 Tablet (Fed) (N=12) | 200-mg LY2940680 Capsule (Fasted) (N=6) | 400-mg LY2940680 Capsule (Fasted) (N=5)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 6 (6) | 3 (3) | 0 (0) | 3 (4) | 3 (3) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0/8 (0) | 0 (0) | 1/19 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/3 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days